CLINICAL TRIAL: NCT02876367
Title: The Clinical Epidemiology of Scrub Typhus in Humans, Chiggers and Rodents
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit (Other); Wellcome Trust (Other); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Other Study IDs: OxTREC no. 48-15
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Scrub Typhus
Keywords: Epidemiology
MeSH Terms: conditions — Scrub Typhus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Group 1: 10 ml of blood will be collected from the participant.
  Group 2: 0.2 ml of blood will be collected from the participant.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute scrub typhus (Group 1): Participants presenting with a fever will be verbally consented for a scrub typhus RDT, using <1ml of blood that is likely to be taken as part of routine clinical assessment. If the RDT tests positive, the patient will be informed about the study and asked to give written informed consent. If they agree to join the study, participants will be asked to give a further blood sample of 10mls (2 teaspoons) for ELISA, PCR and culture testing to confirm the presence of scrub typhus.
- Scrub typhus serosurvey (Group 2): Villagers who are living in an identified scrub typhus environment will be informed about the study and asked to give written informed consent. If they agree to join the study they will be asked to give a finger prick dried blood spot (DBS) test on which scrub typhus ELISA and IFA will be performed.

SUMMARY:
This study to collect and identify rodents and mites across transects through diverse habitats used by the human community from a localised area identified as a scrub typhus 'hot spot'.

DETAILED DESCRIPTION:
Study design:

The project will undertake a detailed investigation of one human community, and its environment, at risk of scrub typhus:

Chiggers, Rodents & Habitat Study:

Transects across diverse habitats determining spatial distribution of species of chiggers and rodents. This will be performed 3x/year.

High-resolution habitat mapping. Comparison of genomes of O. tsutsugamushi detected in different environments, using attempted WGS.

Village Cohort Study:

Follow a cohort of villagers over 2 years screening all febrile patients for scrub typhus and determining seroconversion rates and infecting O. tsutsugamushi genotypes.

Procedures:

* Mites:

Working with ecology/GIS collaborators, the environment of the community will be mapped and transects laid across the diverse habitats used by the community. Free-living mites will be collected with black plastic plates and black cloth21, from soil using Berlese funnels and from rodents. Trombiculid mites will be identified to genus and a subset to species.

DNA will be extracted from individual chiggers, and qPCR screening for O. tsutsugamushi-positivity performed (real-time PCR targeting 47kDa-gene). A proportion of confirmed positives will undergo genotyping by attempted whole-genome sequencing (WGS).

* Rodents:

Rodents will be captured alive along transects and identified in collaboration with University of Montpellier24. All mites will be removed from rodents, the rodents killed and the rodent spleen and liver collected for O. tsutsugamushi qPCR screening. A proportion of O. tsutsugamushi-positive samples will undergo genotyping by attempted WGS or extended MLST analysis.

* Human cohort:

All those in the community (>10 years old) will be approached and asked for consent to participate. All enrolled will have scrub typhus ELISA/IFA (from finger-prick filter paper blood spots) performed every 4 months over 2 years to estimate the rates and dynamics of seroconversion. A brief questionnaire will be administered at each visit to determine whether the participant had a febrile illness in the preceding 4 months.

Patients presenting with a febrile illness to local healthcare facilities will be clinically assessed and an on-site scrub typhus IgM rapid diagnostic test (RDT) performed. RDT positive patients will be recruited into the study, and paired acute/convalescent samples sent to LOMWRU for ELISA, qPCR and BSL3 culture, followed by genotyping by attempted WGS. A questionnaire will be administered to recruited patients to determine symptomatology and vital signs recorded.

Epidemiology & Ecology:

The exact sample collection locations and habitat details will be recorded.

Genomic analyses:

To characterize the relationships between highly diverse O. tsutsugamushi genotypes in multiple strain/genotype-infected hosts a proportion of qPCR positives (approx. 480 samples) will be analysed by whole-genome sequencing at WTCHG in Oxford.

ELIGIBILITY:
Inclusion Criteria:

Acute scrub typhus (Group 1)

1. Presenting with fever >38 C and testing positive by scrub typhus RDT.
2. Male or Female, aged 10 years or above.
3. Participant is willing and able to give informed consent for participation in the study.

Scrub typhus serosurvey (Group 2)

1. Villagers living in an environment in which scrub typhus is known to be present, who are asymptomatic.
2. Male or Female, aged 10 years or above.
3. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

Acute scrub typhus (Group 1)

1. Villagers/patients under 10 years of age.
2. Those unwilling to give written informed consent.

Scrub typhus serosurvey (Group 2)

1. Villagers/patients under 10 years of age.
2. Those unwilling to give written informed consent.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group 1 Male or Female, aged 10 years or above, presenting with a fever
  Group 2 Male or Female, aged 10 years or above, living in an identified scrub typhus environment
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
determine the diversity of O. tsutsugamushi genotypes infecting rodents and mites and link these to their geographical distribution and associated habitat characteristics. | up to 24 months
Correlate the frequency of O. tsutsugamushi in mites and rodents with habitat characteristics, to define interactions between distribution and transmission dynamics. | up to 24 months
Identify key mite vectors and rodent hosts involved in scrub typhus natural history, human infection, and disease virulence | up to 24 months

SECONDARY OUTCOMES:
Determine changes in scrub typhus antibody titres over time and identify acutely infected scrub typhus cases | up to 24 months
Identify human-derived O. tsutsugamushi genotypes to define genomic relationships between human, rodent and mite-derived genotypes. | up to 24 months
Identify putative determinants of human infection/virulence | up to 24 months
To interlink the distribution of O. tsutsugamushi positive mites, rodents and humans with habitat characteristics to propose interventions to reduce the risk of human disease. | up to 24 months

IPD SHARING:
Plan to Share IPD: Yes